CLINICAL TRIAL: NCT04342754
Title: Bilateral Deep Brain Stimulation of Forel's H Field in Tourette's Syndrome: Prospective, Randomized, Crossover, Double-blind Study
Brief Title: Deep Brain Stimulation in Forel's H Field in Tourette's Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rubens Gisbert Cury, Medical Assistant, Movement Disorders Unit. Principal Investigator. MD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3.158.435
Record Dates: First submitted 2020-04-01; First posted 2020-04-13 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Tourette Syndrome
Keywords: DBS; Deep Brain Stimulation; Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Phase 1: Open label phase. All patients are in the ON stimulation condition and will be followed for 6 months.
  Phase 2: Blind phase. All patients will be randomized for ON stimulation or sham stimulation group for 3 months, followed for 1 month of washout and crossover for other group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Brain Stimulation ON (DBS ON) (Experimental): The device will be turned ON
  Interventions: Device: Deep Brain Stimulation (DBS)
- Deep Brain Stimulation OFF (DBS OFF) (Sham Comparator): The device will be turned OFF
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — The device will be ON
  Arms: Deep Brain Stimulation ON (DBS ON)
Device: Sham Stimulation — The device will be OFF
  Arms: Deep Brain Stimulation OFF (DBS OFF)

SUMMARY:
Tourette's Syndrome (TS) is a neurodevelopmental disease characterized tics that start before the age of 18 years. About 5% of cases do not respond to drug treatment and can be classified as refractory and in these cases surgical treatment, with deep brain stimulation, appears as a therapeutic possibility, but with still conflicting results. Our hypothesis is that DBS in Forel's H Field could improve tourette's symptoms, neurological and psychiatric ones.

DETAILED DESCRIPTION:
Sixteen patients with TS will be included in our protocol. The tics must have a negative influence in the quality of life of these patients. Patients will be submitted to a neuronavigation protocol for the precise location of the surgical target. After the surgery all patients will have the device turned ON for 6 months.

After the first 6 months participants will be randomly in two groups, one to stay with device ON or turned OFF at a period of 3 months. After that the groups will cross over for more 3 months. Clinical and video evaluations will be conducted before the surgery, at end of open fase, in the moment of cross over and at end of all.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Tourette's Syndrome diagnosis.
* Age equal to or above 14 years.
* Severe impairment of motor tics (Yale Global Tic Severity Scale ≥ 35/50).
* Patients who are refractory to drug treatment.
* Patients intellectually able to understand and sign the consent form.
* Possibility to adhere to research and periodic medical visits after surgery.

Exclusion Criteria:

* Inability to consent to your participation in the study.
* Patients with non-stabilized psychiatric comorbidities, such as anxiety and depression.
* Concomitant treatment with other experimental drugs.
* Women who are pregnant or breastfeeding.
* Patients undergoing previous neurosurgical procedures for the treatment of Tourette's Syndrome.

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2022-12-27 (Estimated); Study Completion 2023-06-27 (Estimated)

PRIMARY OUTCOMES:
Percent of change in the score of Yale Global Tic Severity Scale (YGTSS) pré and pós stimulation, comparing device On(active) and device OFF (sham) conditions. | month 0: baseline; month 8: end off open label phase. All patients had de device ON for 6 months. month 11: after 3 months of device ON or OFF. month 14: after 3 months of device in opposite situation at evaluation at month 11.
  Assess 5 items: number, frequency, intensity, complexity, interference. Each item is scored for phonic and motor tic symptom by the patient on a 0 to 5 numerical scale. The maximum possible score for these part is 50. Add to that the impairment score, which also has 50 as the maximum score.
  Total Yale Global Tic Severity Scale Score (Total Tic Severity Score + Impairment). The maximum possible score for the total scale is 100.
  Lower scores of YGTSS represents less tics.

SECONDARY OUTCOMES:
Change in psychiatric symptoms - Anxiety | month 0: baseline; month 8: end off open label phase. All patients had de device ON for 6 months. month 11: after 3 months of device ON or OFF. month 14: after 3 months of device in opposite situation at evaluation at month 11.
  To assess the influence of deep brain stimulation on anxiety by comparing specific scales for the quantitative assessment of this symptom. The scale used is Beck Anxiety Inventory (BAI), a self-report measure of anxiety and total score is calculated by finding the sum of the 21 items.
Change in Quality of Life | month 0: baseline; month 8: end off open label phase. All patients had de device ON for 6 months. month 11: after 3 months of device ON or OFF. month 14: after 3 months of device in opposite situation at evaluation at month 11.
  Percent change in the score of Gilles de la Tourette Syndrome - Quality of Life scale (GTS-QOL) comparing baseline, device On and device OFF conditions.
  The GTS-QOL consisted of 27 items and four subscales (psychological, physical, obsessive compulsive and cognitive. Each item is rated across five response options: 'Never', 'Rarely', 'Sometimes', 'Often', 'Always'.
Change in psychiatric symptom - Depression | month 0: baseline; month 8: end off open label phase. All patients had de device ON for 6 months. month 11: after 3 months of device ON or OFF. month 14: after 3 months of device in opposite situation at evaluation at month 11.
  To assess the influence of deep brain stimulation on depression by comparing specific scales for the quantitative assessment of this symptoms. The scale used is the Beck Depression Inventory (BDI), a 21 item self-rated scale that evaluates key symptoms of depression.
Change in psychiatric symptom - obsessive-compulsive disorder | month 0: baseline; month 8: end off open label phase. All patients had de device ON for 6 months. month 11: after 3 months of device ON or OFF. month 14: after 3 months of device in opposite situation at evaluation at month 11.
  To assess the influence of deep brain stimulation on obsessive-compulsive disorder (OCD) by comparing specific scales for the quantitative assessment of this symptoms. The scale used is Yale-Brown Obsessive Compulsive Scale (Y-BOCS), a widely used clinician-rated measure for assessing obsessive-compulsive symptoms.
Change in psychiatric symptom - attention deficit hyperactivity disorder | month 0: baseline; month 8: end off open label phase. All patients had de device ON for 6 months. month 11: after 3 months of device ON or OFF. month 14: after 3 months of device in opposite situation at evaluation at month 11.
  To assess the influence of deep brain stimulation on attention deficit hyperactivity disorder (ADHD) by comparing specific scales for the quantitative assessment of this symptom.The scale used is Adult Self-Report Scale (ASRS-18).
assessment of structural connectivity patterns | month 0: baseline; month 8: end off open label phase. All patients had de device ON for 6 months. month 11: after 3 months of device ON or OFF. month 14: after 3 months of device in opposite situation at evaluation at month 11.
  To assess the variation in the clinical response depending on the pattern of structural connectivity presented by accessing imaging tests of white matter tracts potentially stimulated through ECP targeting the Forel H field.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens G Cury, MD PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided